CLINICAL TRIAL: NCT03119831
Title: A Randomized Controlled Clinical Trial on the Effectiveness of Three Different Mouthrinses, Adjunct to Periodontal Surgery, in Dental Plaque Control and Early Wound Healing
Brief Title: Effectiveness of Three Different Mouthrinses in Dental Plaque Control and Early Wound Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Anastasios M. Gkatzonis, MSc, DDS, MSc, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 269
Record Dates: First submitted 2017-04-09; First posted 2017-04-19 (Actual); Results first posted 2017-07-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Periodontitis; Wound Healing
Keywords: chlorhexidine; alcohol; C31G; Mouthrinses; Early postsurgical wound healing
MeSH Terms: conditions — Periodontitis | interventions — Ethanol; C 31G

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- C31G (Group A) (Experimental): C31G
  Interventions: Drug: C31G
- Alcohol-free Chlorhexidine (Group B) (Experimental): Alcohol-free Chlorhexidine Gluconate 0.12%
  Interventions: Drug: Alcohol-free Chlorhexidine Gluconate 0.12%
- Alcohol-based Chlorhexidine (Group C) (Experimental): Alcohol-based Chlorhexidine Gluconate 0.12%
  Interventions: Drug: Alcohol-based Chlorhexidine Gluconate 0.12%

INTERVENTIONS:
Drug: Alcohol-based Chlorhexidine Gluconate 0.12% — Rinsing with 15ml for one minute twice daily for 14 days
  Arms: Alcohol-based Chlorhexidine (Group C)
Drug: Alcohol-free Chlorhexidine Gluconate 0.12% — Rinsing with 15ml for one minute twice daily for 14 days
  Arms: Alcohol-free Chlorhexidine (Group B)
Drug: C31G — Rinsing with 15ml for one minute twice daily for 14 days
  Arms: C31G (Group A)

SUMMARY:
Aim: This study compared the effectiveness of three different mouthrinses (alcohol and non-alcohol chlorhexidine, alkyl dimethyl glycine / alkyl dimethyl amine oxide - C31G) in plaque control and early wound healing, postoperatively.

Materials and Methods: In this, randomized, double-blind, controlled clinical trial 42 patients were allocated to three groups assigned to two weeks rinsing after periodontal surgery with C31G (group A), alcohol-free chlorhexidine 0.12% (group B) or alcohol-based chlorhexidine 0.12% (group C). At weeks 1 and 2, plaque and early wound healing indices were recorded. At day 14, total bacterial counts were estimated utilizing real - time qPCR. Statistics included linear and generalized linear mixed models.

DETAILED DESCRIPTION:
Materials and Methods

Patients' enrollment and all clinical procedures were conducted at the Department of Periodontology, School of Dentistry, National and Kapodistrian University of Athens, Greece.

Clinical Procedures:

All surgical interventions were conducted by first and third year postgraduate residents. Supragingival debridement and polishing of the operated area was performed immediately before surgery. In cases of residual periodontal pocket elimination / reduction surgeries, intrasulcular incisions followed by papilla preservation incisions at interdental areas were applied. In crown lengthening cases, resective gingival incisions were applied in presence of sufficient width of keratinized tissues (≥ 3mm). Following flap elevation, root surfaces were thoroughly debrided with instruments and ultrasonic devices. Ostectomy / osteoplasty with carbide burs was applied, as deemed appropriate. Buccal and palatal / lingual flaps were fully adapted to each other and sutured together with monofilament slowly resorbable suture. Periodontal dressings were not used. No systemic antibiotics were prescribed. Ibuprofen 400mg, three times daily for 4 days, was suggested immediately after surgical intervention. Smokers were advised to cease smoking for the first postsurgical week. Sutures were removed at 7th postoperative day. During that period no accidental loss of sutures was recorded.

Randomization and allocation concealment:

Subjects were randomly assigned to one of three groups using a computerized assignment procedure (Random Sequence Generator, www.random.org) generated by the examiner A.G. Each subject was given an identical number between 1 and 42. Participants received bottles with one of the three solutions under investigation. Neither patients nor clinicians (surgeons and examiner A.G.) were informed about the identity of mouthrinse administered in each case (double - blind design). Masked bottles were given to participants by a third independent person who was not a dentist (member of Postgraduate Clinic's assistance staff).

Post - surgical maintenance protocol:

During the first 14 postoperative days, participants were instructed to rinse with 15ml of the administered solution for one minute, twice daily.

During the same period, subjects refrained from any mechanical plaque removal at the operated areas.

Intra-examiner reproducibility:

Prior to the beginning of the study, the examiner (A.G.) who performed the measurements was calibrated in order to establish intra - examiner reproducibility. Calibrations were performed with two subjects not included in the study. During post-operative maintenance using 0.12% chlorhexidine, at the 7th postsurgical day, early wound healing index (EHI) and plaque index (PI) were recorded on two separate occasions during the same day, however at least 8 hours apart. Intra-class correlation analysis was used to calculate intra-examiner agreement for repeated measurements. The calibration was accepted if both measurements were similar with a deviation of +/- 10% (intra-class correlation coefficient > 0.9).

Microbiological assessment:

Supragingival dental plaque pooled samples were collected at the 14th postoperative day from both interproximal tooth surfaces respectively to the interdental papilla with the highest EHI value, using curettes. Pooled samples were individually collected in 150μl TE buffer solution. Samples were stored at -80 until processing, which was performed at the Laboratory of Cell and Matrix Pathobiology at the Institute of Biosciences and Applications, National Center for Scientific Research (N.C.S.R.), Athens, Greece. Bacterial genomic DNA was isolated and purified using the PureLink® Genomic DNA Μini Kit, following the Gram (+) bacterial cell lysis manufacturer's protocol. Purified DNA concentrations were determined spectrophotometrically (NanoDrop 1000). Specimens were analyzed using quantitative real time PCR (qPCR) in order to evaluate the total bacterial count in each pooled sample. qPCR was conducted with application of a set of universal primers (forward primer: 5' TCCTACGGGAGGCAGCAGT 3' and reverse primer: 5' GGACTACCAGGGTATCTAATCCTGTT 3', with an amplicon size of 466 base pairs), reported to detect DNA sequences of gene encoding for 16S ribosomal subunit of at least 50 different bacterial species (aerobic and anaerobic Gram positive and Gram negative) and SYBR Green Ι fluorescent probe. Serial dilutions of DNA extract of pure bacterial cultures of Escherichia coli were performed in order to generate a standard curve for the qPCR. Reactions were performed for 40 cycles at 94 °C for 30 sec, 58 °C for 45 sec and 72 °C for 10 min in a Light Cycler 96 qPCR Device. Results were analyzed using the Light Cycler 96 1.1 Software. Total bacterial count of each sample is expressed as total bacterial DNA mass (ng) and bacterial copy numbers (x106).

Sample size calculation:

Sample size was estimated through one-way ANOVA based calculations, assuming that the minimum clinically significant difference is one unit in median EHI values at 14 days between at least one pair of groups. 14 patients for each group were needed for 80% power achievement and for median differences detection in under evaluation parameters among the groups.

Statistical analysis:

Demographic and clinical characteristics of the sample are presented by group in tables containing absolute and relative (%) frequencies for categorical variables and medians and interquartile ranges (Median - IQR) for quantitative variables. Between groups differences in these characteristics were assessed through Fisher's exact tests for categorical variables and Kruskal-Wallis tests for quantitative ones. The distributions of the indices of interest (Early wound healing index - EHI, Plaque index - PI, Plaque area index - PA%) were summarized through medians and IQRs.

Indices' data were analyzed through linear or generalized linear mixed models taking into account the potential correlations between multiple measurements taken on the same individual. In particular, for the analysis of EHI and PI, ordinal logistic regression models were used. For the PA% index, which was a proportion ranging from 0% to 100%, a linear model was used after a logit transformation of the dependent variable. Model selection, including checks for potential interaction effects, for the final multivariable models was based on likelihood ratio tests.

Total microbial count differences among groups or in relation to other sample characteristics were analyzed using linear regression model after log10 transformation. Results are presented as relative differences %.

P-values less than 0.05 were considered statistically significant. All analyses were performed using the statistical package Stata 13.1 (Stata Corp., USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of periodontal pocket elimination / reduction or surgical crown lengthening with or without osseous surgery in one of the following regions: #13-15 or #23-25 or #33-35 or #43-45.
* In cases of pocket elimination / reduction, at least two teeth with ≥ 1 residual periodontal pocket ≥ 5mm and bleeding on probing was mandatory.
* Width of keratinized tissues ≥ 2mm around teeth included in the operated area.
* Cause - related therapy should be completed ≥ 6 weeks before surgical procedure.
* Plaque Index (O'Leary et al. 1972) < 25% and Gingival Bleeding Index (Ainamo and Bay 1975) < 25% in whole dentition should be achieved.

Exclusion Criteria:

* Uncontrolled diabetes mellitus type 1 or 2 (HbA1c > 7%).
* Smoking > 20 cigarettes/day.
* Systemic antimicrobial therapy the last 3 months before the surgical procedure.
* Steroidal or/and non - steroidal anti-inflammatory drug therapy the last 15 days.
* Immunodeficiency or immunosuppressive drug therapy.
* History or current chemotherapy or/and radiation therapy.
* Oral bisphosphonates intake > 3 years or intravenous bisphosphonates therapy.
* Pregnancy or/and breastfeeding.
* Need for osseous graft and/or membrane or any other regenerative material application.
* Furcation involvement of first maxillary premolars and furcation involvement > class I at the mesial entrance of first maxillary molars.
* Missing teeth, fixed partial dentures, removable dentures or orthodontic brackets in the candidate regions for periodontal surgery.

Ages: 34 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phoebus N Madianos, Professor, Study Chair — Department of Periodontology, School of Dentistry, National and Kapodistrian University of Athens, Greece

RESULTS

PARTICIPANT FLOW:
Groups:
- C31G (Group A): C31G
  C31G: Rinsing with 15ml for one minute twice daily for 14 days postoperatively
- Alcohol-free Chlorhexidine (Group B): Alcohol-free Chlorhexidine Gluconate 0.12%
  Alcohol-free Chlorhexidine Gluconate 0.12%: Rinsing with 15ml for one minute twice daily for 14 days postoperatively
- Alcohol-based Chlorhexidine (Group C): Alcohol-based Chlorhexidine Gluconate 0.12%
  Alcohol-based Chlorhexidine Gluconate 0.12%: Rinsing with 15ml for one minute twice daily for 14 days postoperatively
Period: Overall Study
Arm/Group | C31G (Group A) | Alcohol-free Chlorhexidine (Group B) | Alcohol-based Chlorhexidine (Group C)
Started | 14 | 14 | 14
Completed | 14 | 14 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: C31G
  C31G: Rinsing with 15ml for one minute twice daily for 14 days postsurgically
- Group B: Non-alcoholic Chlorhexidine Gluconate 0.12%
  Non-alcoholic Chlorhexidine Gluconate 0.12%: Rinsing with 15ml for one minute twice daily for 14 days postsurgically
- Group C: Alcoholic Chlorhexidine Gluconate 0.12%
  Alcoholic Chlorhexidine Gluconate 0.12%: Rinsing with 15ml for one minute twice daily for 14 days postsurgically
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 14 | 14 | 14 | 42
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [43 to 58] | 52 [49 to 59] | 49 [43 to 55] | 51 [45 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 11 | 28
  Male | 7 | 4 | 3 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Smoking status [Count of Participants; unit: Participants]
  Smoker | 5 | 6 | 5 | 16
  Non - smoker | 8 | 7 | 8 | 23
  Ex - smoker | 1 | 1 | 1 | 3
Surgeon's experience [Count of Participants; unit: Participants]
  Third year postgraduate residents | 11 | 12 | 10 | 33
  First year postgraduate residents | 3 | 2 | 4 | 9
Type of periodontal surgical intervention [Count of Participants; unit: Participants]
  Periodontal flap surgery | 10 | 12 | 8 | 30
  Crown lengthening | 4 | 1 | 5 | 10
  Combination | 0 | 1 | 1 | 2
Tooth area scheduled for surgery [Count of Participants; unit: Participants] — According to FDI World Dental Federation enumeration system:
  * Area #13-17: Maxillary right canine - maxillary right second molar
  * Area #23-27: Maxillary left canine - maxillary left second molar
  * Area #33-37: Mandibular left canine - mandibular left second molar
  * Area #43-47: Mandibular right canine - mandibular right second molar
  Participants
    Area #13-17 | 5 | 4 | 5 | 14
    Area #23-27 | 3 | 2 | 4 | 9
    Area #33-37 | 2 | 3 | 2 | 7
    Area #43-47 | 4 | 5 | 3 | 12
Jaw [Count of Participants; unit: Participants]
  Maxilla | 8 | 6 | 9 | 23
  Mandible | 6 | 8 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Periodontal Soft Tissue Healing Progress Between Baseline (Immediately After Surgery), 7 and 14 Days Postoperatively (Evaluated by Early Wound Healing Index - EHI)
Description: EHI measurements range between 1-5:
  1. = Complete flap closure-no fibrin line in interproximal area.
  2. = Complete flap closure-fibrin line in interproximal area.
  3. = Complete flap closure-fibrin clot in the interproximal area.
  4. = Incomplete flap closure-partial necrosis of interproximal tissue.
  5. = Incomplete flap closure-complete necrosis of the interproximal tissue.
Time Frame: Early Wound Healing Index was recorded at the 7th and 14th postsurgical day
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Group A: C31G
  C31G: Rinsing with 15ml for one minute twice daily for 14 days postoperatively
- Group B: Alcohol-free Chlorhexidine Gluconate 0.12%
  Alcohol-free Chlorhexidine Gluconate 0.12%: Rinsing with 15ml for one minute twice daily for 14 days postoperatively
- Group C: Alcohol-based Chlorhexidine Gluconate 0.12%
  Alcohol-based Chlorhexidine Gluconate 0.12%: Rinsing with 15ml for one minute twice daily for 14 days postoperatively
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 14 | 14
units on a scale
  7 days | 3 [2 to 3] | 3 [2 to 3] | 2 [2 to 3]
  14 days | 2 [1 to 3] | 3 [1 to 4] | 1 [1 to 3]

2. Secondary Outcome: Plaque Index (PI)
Description: PI measurements range between 0-3:
  0 = No plaque
  1. = A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  2. = Moderate accumulation of soft deposits on the tooth and gingival margin which can be seen with the naked eye.
  3. = Abundance of soft matter on the tooth and gingival margin.
Time Frame: PI was recorded 14 days postoperatively
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Group B: Alcohol-free Chlorhexidine Gluconate 0.12%
  Alcohol-free Chlorhexidine Gluconate 0.12%: Rinsing with 15ml for one minute twice daily for 14 days postsurgically
- Group C: Alcohol-based Chlorhexidine Gluconate 0.12%
  Alcohol-based Chlorhexidine Gluconate 0.12%: Rinsing with 15ml for one minute twice daily for 14 days postsurgically
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 14 | 14
units on a scale | 2 [1 to 3] | 2 [1 to 2] | 1 [1 to 1]

3. Secondary Outcome: Plaque Area Index (PA%)
Description: Assessment of the accumulation of dental plaque at buccal tooth surfaces between baseline (immediately before surgery), 7 and 14 days postoperatively. PA% referred at the percentage of the total buccal surface area of the included teeth covered by dental plaque. PA% values range between 0-100%
Time Frame: PA% was recorded at the 7th and 14th postoperative day
Measure: Median (Inter-Quartile Range); unit: percentage of buccal surface area
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 14 | 14
percentage of buccal surface area
  7 days | 22.8 [14.2 to 46.7] | 20.6 [6.3 to 32.2] | 11.2 [6 to 16.5]
  14 days | 32.5 [17.2 to 44.1] | 14.9 [7.6 to 28.6] | 11.2 [4.6 to 29]

4. Other Pre Specified Outcome: Total Bacterial Counts (TBC)
Description: Levels of bacterial counts, expressed in total bacterial DNA mass (ng) and total number of bacteria. TBC was evaluated by real-time Polymerase Chain Reaction (PCR).
Time Frame: Plaque samples were collected at the 14th postsurgical day.
Population: The inconsistency between the overall number of participants analyzed and the numbers provided in the rows in the participant flow module is due to the fact that there were no microbiological data from three patients in Group B and from another three participants in Group C, because their pooled plaque samples were destroyed during processing.
Measure: Median (Inter-Quartile Range); unit: log10 of copy numbers of bacterial DNA
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 14 | 11 | 11
log10 of copy numbers of bacterial DNA | 7.584 [7.421 to 7.835] | 7.683 [7.425 to 8.046] | 6.480 [5.869 to 7.065]

ADVERSE EVENTS:
Arm/Group | Group A | Group B | Group C
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes